CLINICAL TRIAL: NCT07349667
Title: Hypnotherapy for Needle-related Procedural Pain and Anxiety Management in a Pediatric Setting: A Randomized Controlled Trial
Brief Title: Hypnotherapy for Needle-related Procedural Pain and Anxiety Management in a Pediatric Setting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Claus Sixtus Jensen, Associate professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0097327
Record Dates: First submitted 2025-09-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Juvenile; Arthritis, Juvenile Idiopathic; Lupus Erythematosus, Systemic; Dermatomyositis, Juvenile
Keywords: Hypnotherapy; pediatric; needle fear
MeSH Terms: conditions — Arthritis, Juvenile; Lupus Erythematosus, Systemic; Dermatomyositis; Iatrophobia | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnotherapy (Other): Childrenin the intervention group will receive hypnotherapy sessions conducted by one of two trained and certified hypnotherapists. The sessions will be tailored to the child's age and understanding
  Interventions: Other: Hypnotherapy
- Control group (No Intervention): Children in the control group will receive standard care for pain management during medical procedures.

INTERVENTIONS:
Other: Hypnotherapy — The hypnotherapy session will be individualized to the particular child. The nurse performing the hypnotherapy session will ask the child a few basic questions about his/her favorite place or activity. If the child do not have any suggestions the nurse will suggest an age-appropriate activity to daydream about, such as making a snowman for a six year-old or skiing for an adolescent, and then suggest a hypnotic "daydream" about that place or activity. Most inductions for older children (ages approximately 9-15) included a few slow, deep breaths and/or some progressive relaxation, such as muscle relaxation or the suggestion of a "warm, comfortable feeling" flowing up the body from the feet to the head. Younger children, unless they expressed an interest in deep breathing or relaxation, will typically asked simply to imagine themselves arriving at their favorite place and/or beginning their favorite activity.
  Arms: Hypnotherapy

SUMMARY:
The proposed study aims to evaluate the effectiveness of hypnotherapy as a non-pharmacological intervention for managing pain and anxiety during needle-related medical procedures in children aged 5 to 17 years. This research addresses a significant gap in pediatric healthcare, where painful procedures often induce distress and long-term anxiety, leading to avoidance of necessary medical care. Conventional pain management strategies primarily rely on pharmacological methods, which may pose risks and side effects. Thus, exploring safe and effective alternatives, such as hypnotherapy, is crucial.The target group for this randomized controlled trial includes children scheduled for painful procedures, such as injections or blood sampling. Participants will be randomly assigned to either the hypnotherapy group, receiving tailored sessions conducted by trained hypnotherapists, or the standard of care group, which will involve conventional pain management techniques. The study will assess primary outcomes, including anxiety levels and pain perception, before, during, and after the procedures using validated scales.

Key activities of the project include conducting individualized hypnotherapy sessions, monitoring anxiety and pain levels through structured assessments, and analyzing the data to determine the effectiveness and feasibility of hypnotherapy. Secondary objectives will explore potential long-term benefits and safety concerns associated with hypnotherapy. If successful, this study could significantly enhance pediatric pain management practices, reduce reliance on pharmacological interventions, and improve the overall healthcare experience for children. The findings may also inform broader healthcare policies regarding non-pharmacological pain management strategies in pediatric settings.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 18 years
* Scheduled for a painful medical procedure (injections or blood sampling)
* Informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Children with a history of psychiatric disorders or cognitive impairment
* Children unable to understand and participate in hypnotherapy sessions
* Any contraindication to hypnotherapy
* Children with diagnosed cancer

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Level of anxiety before, during and after the medical procedure and pain intensity before, during and after the medical procedure. | pre-procedure, periprocedurally and immediately after the procedure
  Anxiety will be measure using Modified Yale Preoperative Anxiety Scale. The instrument contains 27 items in five categories indicating anxiety in children (activity, emotional expressivity, state of arousal, vocalization, and use of parents). Scores range from 22 to 100; higher scores indicate higher levels of anxiety.

SECONDARY OUTCOMES:
Generalized anxiety. | Immediately after the procedure
  Spence Children's Anxiety Scale. The Spence Children's Anxiety Scale - Child Version (SCAS-Child) is a 44-item self-report measure, with responses recorded on a 4-point scale ranging from 0 (never) to 3 (always), designed to assess anxiety symptoms in children aged 8-15 years. Built upon contemporary diagnostic frameworks, the SCAS-Child evaluates six distinct domains of anxiety that align with clinical diagnostic categories. A higher score on the Spence Children's Anxiety Scale (SCAS) indicates a greater severity and number of anxiety symptoms, suggesting the child experiences more significant anxiety, which can be further broken down into subscales for specific fears like separation anxiety, social phobia, or panic.
Adverse events related to hypnotherapy | Immediately after the procedure
  Adverse events related to hypnotherapy. Will be evaluated by asking patients to rate nausea and dizziness on a self-constructed 4-point scale (range 0-3; 0, no nausea/dizziness at all; 3, severely nauseous/dizzy).
The time spend on the total procedure | from start to end of procedure
  time spend on the intervention and the needle-related procedure.
Heartrate | pre-procedure, periprocedurally and immediately after the procedure
  Heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study cannot be shared. As a single-center study with a small cohort, participants could potentially be re-identified even after anonymization. Sharing the data would therefore risk exposing sensitive personal or health information.